CLINICAL TRIAL: NCT05639309
Title: Pilot Study to Evaluate the Usefulness of Liver Regional Oxygen Saturation (RSO2) in Preterm Patent Ductus Arteriosus
Brief Title: Liver Regional Oxygen Saturation in Preterm Patent Ductus Arteriosus
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sook Kyung Yum, Dr. Sook Kyung Yum, Seoul St. Mary's Hospital
Other Study IDs: KC22ONSI0820
Record Dates: First submitted 2022-11-22; First posted 2022-12-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Patent Ductus Arteriosus; Circulation; Newborn Morbidity; Premature Birth
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Case (hemodynamically significant patent ductus arteriosus): Hemodynamically significant patent ductus arteriosus (hsPDA) diagnosed by echocardiographic criteria including pulsatile left-to-right shunt through patent ductus arteriosus, enlarged left atrium and/or left ventricle, increased left pulmonary artery velocity, absent or reversed end-diastolic flow of anterior cerebral artery and/or renal artery
  Interventions: Device: near-infrared spectroscopy based cerebral/somatic oximeter system (INVOS™ system manufactured by Medtronics)
- Control (no hemodynamically significant patent ductus arteriosus): no hsPDA based on the same echocardiographic criteria described for the Case group
  Interventions: Device: near-infrared spectroscopy based cerebral/somatic oximeter system (INVOS™ system manufactured by Medtronics)

INTERVENTIONS:
Device: near-infrared spectroscopy based cerebral/somatic oximeter system (INVOS™ system manufactured by Medtronics) — regional oxygen saturation measurement

SUMMARY:
This study evaluates the usefulness of liver perfusion and oxygenation status using regional oxygen saturation (RSO2) values obtained via near-infrared spectroscopy in assessing the hemodynamical significance of patent ductus arteriosus in preterm infants.

DETAILED DESCRIPTION:
The usefulness of cerebral and renal regional oxygen saturation (RSO2) values for assessing hemodynamically significant patent ductus arteriosus (hsPDA) has been described previously. Meanwhile, autoregulation of the splanchnic organs' perfusion is less developed compared to the cerebral and renal system, which makes the splanchnic bed more prone to perfusion decrease and ischemia in cases of volume depletion or poor circulation. If RSO2 is measure in the liver, the solid organ reflecting the splanchnic bed perfusion status, hsPDA may be more readily identified than when only cerebral and/or renal RSO2 is monitored.

This study aims to evaluate the usefulness of liver RSO2 measurement in assessing the hemodynamical significance of patent ductus arteriosus in preterm infants, in comparison to cerebral and renal RSO2.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth less than 32 weeks
* Birthweight less than 1,500 grams

Exclusion Criteria:

* Major congenital anomaly
* chromosomal / genetic anomaly

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born at less than 32 weeks' gestation and/or 1,500 grams at birth, who accepts informed consent from the their legal guardians (parents) will be included. Those with major congenital anomaly or genetic abnormality who are at high risk for adverse outcome and compensated circulatory status will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Day 2 liver regional oxygen saturation | 48 to 72 hours of birth
  regional oxygen saturation of liver obtained from near-infrared spectroscopy (%)
Day 7 liver regional oxygen saturation | 7 (±2) days after birth
  regional oxygen saturation of liver obtained from near-infrared spectroscopy (%)
Day 14 liver regional oxygen saturation | 14 (±3) days after birth
  regional oxygen saturation of liver obtained from near-infrared spectroscopy (%)

SECONDARY OUTCOMES:
PDA liver regional oxygen saturation | When hemodynamically significant patent ductus arteriosus is clinically suspected by the attending physician, up to 28th day of life
  regional oxygen saturation of liver obtained from near-infrared spectroscopy (%)

OTHER OUTCOMES:
Day 2 cerebral regional oxygen saturation | 48 to 72 hours of birth
  regional oxygen saturation of brain obtained from near-infrared spectroscopy (%)
Day 7 cerebral regional oxygen saturation | 7 (±2) days after birth
  regional oxygen saturation of brain obtained from near-infrared spectroscopy (%)
Day 14 cerebral regional oxygen saturation | 14 (±3) days after birth
  regional oxygen saturation of brain obtained from near-infrared spectroscopy (%)
PDA cerebral regional oxygen saturation | When hemodynamically significant patent ductus arteriosus is clinically suspected by the attending physician, , up to 28th day of life
  regional oxygen saturation of brain obtained from near-infrared spectroscopy (%)
Day 2 renal regional oxygen saturation | 48 to 72 hours of birth
  regional oxygen saturation of kidney obtained from near-infrared spectroscopy (%)
Day 7 renal regional oxygen saturation | 7 (±2) days after birth
  regional oxygen saturation of kidney obtained from near-infrared spectroscopy (%)
Day 14 renal regional oxygen saturation | 14 (±3) days after birth
  regional oxygen saturation of kidney obtained from near-infrared spectroscopy (%)
PDA renal regional oxygen saturation | When hemodynamically significant patent ductus arteriosus is clinically suspected by the attending physician, , up to 28th day of life
  regional oxygen saturation of kidney obtained from near-infrared spectroscopy (%)

CONTACTS AND LOCATIONS:
Overall Officials: Sook Kyung Yum, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic Univeristy of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seocho-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No